CLINICAL TRIAL: NCT00892125
Title: Evaluation of the Effect of Carbamazepine on the Steady-state Pharmacokinetics of Paliperidone Extended Release in Clinically Stable Subjects With Schizophrenia or Bipolar I Disorder
Brief Title: A Study of the Effect of Carbamazepine on the Pharmacokinetics of Paliperidone Extended Release (ER) in Patients With Schizophrenia or Bipolar I Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR011440
Record Dates: First submitted 2008-11-20; First posted 2009-05-04 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: Schizophrenia; Bipolar I disorder; mood disorders; antipsychotic drugs; enzyme inducer; Paliperidone ER
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Mood Disorders | interventions — Paliperidone Palmitate; Carbamazepine

INTERVENTIONS:
Drug: paliperidone ER; Carbamazepine

SUMMARY:
The purposes of this study are to evaluate the effects of a potent metabolic enzyme inducer, carbamazepine, on the steady-state pharmacokinetics of orally administered paliperidone ER and to evaluate the safety and tolerability of the treatments in clinically stable patients with a diagnosis of schizophrenia or bipolar I disorder.

DETAILED DESCRIPTION:
The current study is designed as an open-label, multiple-center, multiple-dose, 2 treatment, 2 period sequential drug interaction study. It consists of 3 phases: a screening phase beginning within 21 days before the first study drug administration; an open label treatment phase consisting of 2 treatment periods (Period 1 and Period 2), during which patients will receive multiple oral doses of 6-mg paliperidone ER alone or in combination with multiple oral doses of carbamazepine, and end of study evaluations upon completion of all the study procedures in Period 2 or at early withdrawal. There is no washout period between treatment periods. Given the potential concomitant use of carbamazepine with antipsychotics, such as paliperidone ER, in the treatment of schizophrenia or bipolar I disorder, this study is designed to investigate the effect of carbamazepine on the steady-state pharmacokinetics of paliperidone ER. Safety and tolerability will be monitored throughout the study.. Period 1: 6 mg paliperidone ER once daily from Day 1 through Day 7, route oral; Period 2: 6 mg paliperidone ER once daily and carbamazepine 200 mg twice daily from Day 8 through Day 28, route oral.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia of any subtype (295.10
* 295.20
* 295.30
* 295.60
* 295.90) or bipolar I disorder (296.0x, 296.4x, 296.5x, 296.6x or 296.7), according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)
* Clinically stable with no psychiatric hospitalization or change in existing mood stabilizers, antipsychotic, or anti-manic drugs for 3 months before screening. A reduction in the dose of existing medication is acceptable if the subject remained clinically stable throughout the 3 month period. In addition, an increase or decrease in the dose of a mood stabilizer on the basis of therapeutic drug monitoring or the substitution of a specific mood stabilizer, antipsychotic, or anti-manic drug for another because of poor tolerability will be allowed within 3 months before screening
* Have a CGI-S score of 3 or less at baseline and at screening
* Body mass index (BMI, weight [kg]/height [m2]) of 18 to 35 kg/m2, inclusive
* Have a supine (after 5 minutes rest) blood pressure between 100 and 140 mmHg systolic, inclusive, and 50 and 90 mmHg diastolic, inclusive
* Apart from the above-mentioned diagnosis, otherwise healthy on the basis of a prestudy physical examination, medical history, 12-lead ECG, and the laboratory results of serum chemistry, hematology, and urinalysis performed within 21 days before the first dose. For renal function tests, the values must be within the normal laboratory reference ranges
* Women must be postmenopausal for at least 2 years, surgically sterile, abstinent, or practicing or agree to practice an effective method of birth control if they are sexually active before entry and throughout the study (effective methods of birth control include intrauterine devices, double-barrier method, and male partner sterilization). Prescription hormonal contraceptives must be used in combination with another method of birth control (e.g., double-barrier method) throughout the study. Women of childbearing potential must have a negative serum pregnancy test result at screening, and a negative urine test at baseline (Day 1).

Exclusion Criteria:

* Diagnosis of schizoaffective disorder (295.70) according to the DSM-IV
* Meet DSM-IV criteria for rapid cycling
* DSM-IV diagnosis of alcohol or substance dependence, with the exception of nicotine or caffeine dependence, within 12 months before screening. Intermittent substance abuse in the months before screening will not be exclusionary, depending upon the clinical judgment of the investigator, with the exception of barbiturates
* Acute substance abuse, as evidenced by a positive urine drug screen at screening or baseline (Day 1)
* Positive alcohol test at screening or baseline (Day 1)
* Current suicidal ideation or violent tendencies at the time of screening
* Involuntarily-hospitalized subjects
* Moderate or severe tardive dyskinesia at the time of screening
* History of neuroleptic malignant syndrome
* History of bone marrow depression or acute intermittent porphyria
* History of or a positive result at screening for any of the serology tests (hepatitis B, C, and human immunodeficiency virus [HIV])
* History or presence of any relevant cardiovascular (including myocardial infarct or cardiac arrhythmia), respiratory, neurologic (including seizures), renal, hepatic, gastrointestinal (including surgeries, severe gastrointestinal narrowing, and malabsorption problems), endocrine, hematologic, or immunologic disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2006-09; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
to evaluate the effects of a potent enzyme inducer, carbamazepine, on the steady-state pharmacokinetics of orally administered paliperidone ER

SECONDARY OUTCOMES:
to evaluate the safety and tolerability of the treatments in clinically stable patients with a diagnosis of schizophrenia or bipolar I disorder

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the effect of carbamazepine on the pharmacokinetics of paliperidone extended release (ER) in patients with schizophrenia or bipolar I disorder. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=734&filename=CR011440_CSR.pdf